CLINICAL TRIAL: NCT05721157
Title: Osteoporotic Precisely Screening Using Chest Radiograph and Artificial Neural Network (OPSCAN): a Randomized Controlled Trial
Brief Title: Osteoporotic Precisely Screening Using Chest Radiograph and Artificial Neural Network (OPSCAN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Chin Lin, Associate Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NDMC2023001
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Osteoporosis; Osteoporotic Fractures
MeSH Terms: conditions — Osteoporosis; Osteoporotic Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients randomized to intervention will have access to the screening tool.
  Interventions: Other: AI-enabled Chest X-ray-based Screening Tool
- Control (No Intervention): Patients randomized to control will continue routine practice.

INTERVENTIONS:
Other: AI-enabled Chest X-ray-based Screening Tool — Primary care clinicians in the intervention group had access to the report, which displayed whether the AI-Chest X-ray result was positive or negative.The system will send a message to corresponding physicians if positive finding.
  Arms: Intervention

SUMMARY:
Artificial Intelligence-assisted Diagnosis and Prognostication in Osteoporosis Using Chest X-ray

ELIGIBILITY:
Inclusion Criteria:

* Patients recieved at least 1 chest X-ray examination in 2022
* More than 66% chest X-ray identified as high risk of osteoporosis by AI-CXR

Exclusion Criteria:

* Patients with history of at least 1 dual energy x-ray absorptiometry (DXA)
* Patients with history of osteoporosis or osteoportic fracture
* Patients recieved prescription anti-osteoporotic treatment (excluding vitamin D or calcium)
* Patients died before 01 Jan 2023

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4912 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
newly diagnosed with osteoporosis | Within 180 days
  After performing an chest X-ray, the osteoporosis was followed.

SECONDARY OUTCOMES:
initiation of DXA examination | Within 180 days
  After performing an chest X-ray, the osteoporosis was followed.
initiation of anti-osteoporotic treatment | Within 180 days
  After performing an chest X-ray, the osteoporosis was followed.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-service general hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No